CLINICAL TRIAL: NCT01125241
Title: A Study to Evaluate the Efficacy and Safety of Add-on Therapy of Wuling Capsule in Epilepsy Patients With Depression: a Muli-center, Randomized, Double-blinded, Placebo-controlled Superiority Clinical Trial
Brief Title: A Study to Evaluate the Efficacy and Safety of Add-on Therapy of Wuling Capsule in Epilepsy Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Wu Mengchao Medical Foundation (Unknown); Shanghai Ankang Pharmaceutical Co.,LTD (Unknown)
Responsible Party: Principal Investigator, Weifeng Peng, neurology department, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WL-2010
Record Dates: First submitted 2010-04-26; First posted 2010-05-18 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Epilepsy; Depression
Keywords: wuling capsule; epilepsy; depression; superiority clinical research
MeSH Terms: conditions — Epilepsy; Depression | interventions — wuling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wuling capsule (Experimental)
  Interventions: Drug: wuling capsule
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo of wuling capsule

INTERVENTIONS:
Drug: wuling capsule — orally, three tablets each time,three times a day
  Arms: Wuling capsule
Drug: placebo of wuling capsule — orally, three tablets each time and three times a day
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the effects of add-on therapy of wuling capsule on depressive symptoms in patients with comorbidity of epilepsy and depression, to evaluate its influences on the frequency and severity of seizures, and to observe its effects on patients' sleeping condition, quality of life.

DETAILED DESCRIPTION:
The phenomenon of epileptic patients who have psychiatric disorders is very common, of which the prevalence of depression is the highest and depression is also an independent risk factor affecting epileptic patients' quality of life. Due to some social factors, non-typical clinical symptoms and limited therapeutic methods(tricyclic antidepressants, lithium chloride and 5-serotonin uptake inhibitors may all have risks of lowing threshold of seizures), epileptic patients with depression are usually not be recognized and treated properly. Wuling capsule has been used in therapy of insomnia, nervous breakdowns and a previous small sample clinical trial revealed that it could improve mood disorders of epileptic patients and hadn't affected severity of seizures (not published). Therefore a multi-center, randomized, double-blinded and placebo-controlled superiority clinical trial will be carried out to determine the effects of add-on therapy of wuling capsule on depressive symptoms in patients with epilepsy, to evaluate its influences on the frequency and severity of seizures, and to observe its effects on patients' sleeping condition, quality of life.

ELIGIBILITY:
Inclusion Criteria:

Subjects for this study will meet the following criteria:

1. Age greater than or equal to 18 years.
2. Must be in accordance with the diagnostic criteria of epilepsy and have taken antiepileptic drugs regularly at least for 6 months, which will not be changed recently. The duration to the latest seizure must be longer than 24 hours.
3. Score of a 17 item Hamilton Depression is greater than or equal to 17 and depressive symptoms have lasted for at least 2 weeks.
4. Haven't taken any anti-anxiety, anti-depressant and anti-psychotic drugs in recent 2 weeks.
5. Must sign the informed consent form.

Exclusion Criteria:

1. Now accepting or have accepted other drugs clinical trial in the last month.
2. History of serious psychiatric illness other than depression.
3. Having suicide ideas or suicide behaviors.
4. Progressive illness of central nervous system, such as degenerative disease or tumor.
5. History of serious cardiac or pulmonary disease, hepatic and renal dysfunction, and malignant tumors.
6. The value of ALT or AST is higher than 1.5 times normal range, or the number of white blood cells is less than 2500/ul, or the number of neutrophil granulocyte is less than 1000/ul.
7. During pregnant or lactation period.
8. The person who is disabled or mentally disabled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
symptoms of depression using the 17-item Hamilton Depression Rating Scale (HDRS) | 3 months

SECONDARY OUTCOMES:
the frequency of seizures using diary | 3 months
the severity of seizures using the National Hospital Seizure Severity Scale(NHS3) | 3 months
the sleeping condition using Pittsburgh Sleep Quality Index (PSQI) | 3 months
the quality of life using Quality of Life in Epilepsy (QOLIE-31) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang Xin, MD, Principal Investigator — Fudan University
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, China, Beijing, Beijing Municipality
  - the Second Affiliated Hospital of Guangzhou Medical College, Guangzhou, China, Guangzhou, Guangdong
  - Shanghai Fifth People's Hospital, Shanghai, Shanghai Municipality
  - Department of Neurology, Zhongshan Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality
  - Department of Neurology, Huashan Hospital, Fudan University, Shanghai, China, Shanghai, Shanghai Municipality
  - Department of Neurology, Renji Hospital, Shanghai Jiaotong University, Shanghai, China, Shanghai, Shanghai Municipality
  - the Sixth People's Hospital of Shanghai Jiaotong University，Shanghai,China, Shanghai, Shanghai Municipality
  - Department of Neurology, Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - the First Municipal Hospital of Guangzhou, Guangzhou